CLINICAL TRIAL: NCT06124677
Title: Anatomical and Visual Outcomes Following a Single Injection of Intravitreal Faricimab in Patients With Neovascular Age-related Macular Degeneration and Persisting Fluid Despite Frequent Aflibercept Treatments
Brief Title: Single Injection of Faricimab for nAMD With Persisting Fluid Despite Frequent Aflibercept Treatments
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Staff Specialist, Rigshospitalet, Denmark
Other Study IDs: VAB1SHOT
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients who received intravitreal faricimab injections between May and September, in 2023. and conform the inclusion/exclusion criteria.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — The Injections were performed according to local standard protocol, that included the use of 2-3 drops of topical tetracaine anesthesia, use of eye speculum, topical 5% povidone-iodine disinfection, a 30G-needle, injection site 3.5 mm posterior from the limbus marked by calipers in supertemporal or inferotemporal quadrants, a sterile cotton tip tamponade at the site of injection after removal of the needle, and no post-procedure antibiotics.
  Other Names: Vabysmo (6 mg, 0.05 ml)

SUMMARY:
The goal of this retrospective single-center chat review is to establish the efficacy and safety of a single dose of intravitreal faricimab (Vabysmo®) injection in patients with neovascular age-related macular degeneration (AMD), who were previously treated with aflibercept (Eylea®) and had persisting intraretinal or subretinal fluid despite frequent treatments.

ELIGIBILITY:
Inclusion criteria

* Presence of neovascular age-related macular degeneration (AMD) in the study eye
* >50 years of age
* Previous intravitreal anti-VEGF treatment with aflibercept (Eylea®) or with aflibercept and ranibizumab (Lucentis®) in the study eye
* Minimum of 6 monthly aflibercept injections
* Persisting intraretinal or subretinal fluid or both, despite at least 3 consecutive monthly aflibercept injections in the study eye before switching to faricimab

Exclusion criteria

* Neovascular conditions other than AMD (e.g., choroidal neovascularisation due to other causes) or co-existence of other retinal disease in the study eye
* Significant optical media opacities that would result in poor imaging quality on OCT scans in the study eye
* Intraocular surgery in the study eye 3 months before or within 1 month after the treatment switch

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular age-related macular degeneration (AMD)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients responding to the treatment switch | 4 weeks
  Defined as reduction or disappearance of the intra- or subretinal fluid at 4 weeks following a single injection of faricimab

SECONDARY OUTCOMES:
Durability of a single injection in cases of favorable treatment response without residual fluid | Up to 16 weeks
  Time of reappearance of the fluid
Differences in patient characteristics between individuals responding and not responding to faricimab | 4 weeks
Changes in visual acuity after the treatment switch | 4 weeks
Changes in central retinal thickness after the treatment switch | 4 weeks
  Measured on optical coherence tomography (OCT) scans
Changes in pigment epithelium detachment (PED) height after the treatment switch | 4 weeks
  Measured on optical coherence tomography (OCT) scans

OTHER OUTCOMES:
Frequency of ocular and systemic adverse events | 4 weeks
  As safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, MD, PhD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Miklos Schneider, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schneider M, Bjerager J, Hodzic-Hadzibegovic D, Klefter ON, Subhi Y, Hajari J. Short-term outcomes of treatment switch to faricimab in patients with aflibercept-resistant neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2024 Jul;262(7):2153-2162. doi: 10.1007/s00417-024-06421-0. Epub 2024 Feb 28. PMID 38416237